CLINICAL TRIAL: NCT03623061
Title: A Clinical Study to Define Precision, Accuracy, and Comparability of Results From a Novel Point of Care Fibrinogen Assay (F-Point), Compared to an Industry Standard
Brief Title: F-Point Validation Study
Acronym: F-Point
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Dublin City University (Other); Enterprise Ireland (Other Government)
Responsible Party: Sponsor
Other Study IDs: FPoint-V1-0418
Record Dates: First submitted 2018-06-21; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Low Fibrinogen
MeSH Terms: conditions — Afibrinogenemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low Fibrinogen Level: Anonymised low fibrinogen adult samples from the laboratory (Low fibrinogen concentrations). Samples to be tested on the F-Point device and standard Clauss Fibrinogen assay.
  Interventions: Diagnostic Test: F-Point
- Normal Fibrinogen Level: Healthy non pregnant females presenting for elective gynaecology surgery (Normal non pregnant fibrinogen concentrations) Samples to be tested on the F-Point device and standard Clauss Fibrinogen assay.
  Interventions: Diagnostic Test: F-Point
- High Fibrinogen Level: Healthy pregnant females presenting for elective caesarean section (Normal term pregnancy fibrinogen levels) Samples to be tested on the F-Point device and standard Clauss Fibrinogen assay.
  Interventions: Diagnostic Test: F-Point

INTERVENTIONS:
Diagnostic Test: F-Point — F-Point (point of care in vitro diagnostic device for measuring plasma fibrinogen concentration)

SUMMARY:
The F-Point investigation is an open label, single centre prospective observational study in 3 cohorts of patients, one with low fibrinogen concentration, one with normal fibrinogen concentration, and one with high fibrinogen concentration To show statistical agreement between the fibrinogen level as recorded by the standard lab Clauss fibrinogen, and the fibrinogen level as recorded by the novel F-Point device.

DETAILED DESCRIPTION:
The area to be investigated is the measurement of blood fibrinogen concentration. The aim is to develop a device which can give a fibrinogen level rapidly and accurately, in order to allow decision making quickly in emergency haemorrhage situations.

Postpartum hemorrhage (PPH) is one of the leading causes of maternal mortality and morbidity throughout the world and is accountable for 27.1% of maternal deaths worldwide according to a recent WHO systematic analysis.1 The confidential enquiry into maternal deaths and morbidity 2012 - 2014 describes 13 deaths from maternal haemorrhage.2 Fibrinogen is an component of the coagulation cascade. It is the principal factor for the final stage of clot formation. The fibrinogen level increases during pregnancy from the first through to third trimester.3 During a PPH this level decreases rapidly, influenced by two principal mechanisms, the loss of the blood itself and the consumption of coagulation factors associated with coagulation activation. Fibrinogen level below 2g/L in the early phase of PPH correlates with subsequent development of severe PPH.4 The conventional laboratory tests (Clauss, PT-derived) are time consuming, and workload intensive for laboratory staff. This has implications in terms of decision making in a rapidly changing clinical environment during a massive PPH. A point of care test, with more rapidly available results at the patient location should improve the speed of decision making based on individual patient data. The focus of this study is to validate the fibrinogen concentration as measured by the F-point device compared to the laboratory standard Clauss fibrinogen. The F-Point is second generation POC device that is compatible with deployment within the emergency room or operating theater. By having rapid access to fibrinogen concentration results, early and individualized treatment can be implemented with the aim of improving patient outcomes, with a possible decrease in unnecessary administration of fibrinogen.

We aim to show equivalent performance between the F-Point device in 3 populations.

1. Healthy non-pregnant females presenting for elective gynaecology surgery
2. Healthy pregnant females presenting for elective caesarean section
3. Anonymised low fibrinogen adult samples from the laboratory

These 3 populations have been chosen to demonstrate device performance in:

1. Normal non-pregnant fibrinogen concentrations
2. Normal term pregnancy fibrinogen levels
3. Low fibrinogen concentrations By demonstrating equivalent and acceptable performance at these 3 fibrinogen concentration ranges, we would expect to show performance of the device to be acceptable for clinical use across the spectrum of patients presenting to maternity hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the clinical investigation.
* Female, aged 18 years or above.
* Able (in the Investigators opinion) and willing to comply with all clinical investigation requirements.
* Presenting for Group 1: Elective Caesarean section Group 2: Elective gynaecological procedure
* Group 3 will consist of anonymous patient samples

Exclusion Criteria:

* Patients on any antiplatelet or anticoagulant medications

  o Patients prescribed subcutaneous low molecular weight heparin medications are permitted to enrol, provided the timing of sampling is outside of 24 hours after the last dose of the medication.
* Any patient with a known thrombophilia or a known haemophilia.
* Any patient with a known dysfibrinogenaemia except in the anonymous low fibrinogen group
* Patients with a known malignancy or autoimmune condition affecting blood clotting
* A personal history of easy bruising strongly suggestive of a blood clotting disorder
* Any reason, in the opinion of the investigator that would make the subject unsuitable for participation

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Group 1: Elective Caesarean section Group 2: Elective gynaecological procedure
  •Group 3 will consist of anonymous patient samples
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of Fibrinogen concentration | Within 2 hours of blood drawn
  To demonstrate equivalent performance between a novel point of care device, the F-point, when compared to the laboratory Clauss assay for measuring fibrinogen concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Thornton, Principal Investigator — Rotunda Hospital
Locations (1):
- Obstetrics & Gynaecology, The Rotunda Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Result] Gong JM, Shen Y, He YX. Reference Intervals of Routine Coagulation Assays During the Pregnancy and Puerperium Period. J Clin Lab Anal. 2016 Nov;30(6):912-917. doi: 10.1002/jcla.21956. Epub 2016 Apr 7. PMID 27061783
- [Result] Charbit B, Mandelbrot L, Samain E, Baron G, Haddaoui B, Keita H, Sibony O, Mahieu-Caputo D, Hurtaud-Roux MF, Huisse MG, Denninger MH, de Prost D; PPH Study Group. The decrease of fibrinogen is an early predictor of the severity of postpartum hemorrhage. J Thromb Haemost. 2007 Feb;5(2):266-73. doi: 10.1111/j.1538-7836.2007.02297.x. Epub 2006 Nov 6. PMID 17087729